CLINICAL TRIAL: NCT04574141
Title: Randomized, Open-label Bioavailability Study of the Kinetics of Plasma, Urinary and Salivary Concentrations of Melatonin and 6-sulfatoxymelatonin Subsequent to the Consumption of Melatonin-rich Food Supplements With Different Galenic Forms
Brief Title: Kinetic of Melatonin Subsequent to the Consumption of Melatonin-rich Food Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PiLeJe (Industry)
Responsible Party: Sponsor
Organization: Larena SAS (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pil-Clin-Melat-020
Record Dates: First submitted 2020-07-27; First posted 2020-10-05 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Melatonin Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spray before tablet (Experimental)
  Interventions: Dietary Supplement: a prolonged release tablet and a spray containing melatonin
- tablet before spray (Experimental)
  Interventions: Dietary Supplement: a prolonged release tablet and a spray containing melatonin

INTERVENTIONS:
Dietary Supplement: a prolonged release tablet and a spray containing melatonin — prolonged release tablet is dosed at 1.9mg and spray is dosed at 1mg for 2 oral sprays.

SUMMARY:
This study is conducted to clinically document the melatonin bioavailability of two dietary supplements containing melatonin : one prolonged release tablet dosed at 1.9mg and one spray dosed at 1mg for 2 oral sprays.

ELIGIBILITY:
Inclusion Criteria:

* Male between the ages of 18 and 45,
* In good general health, i.e., free of chronic conditions and not taking medication at the time of inclusion and/or long-term,
* Over 70 kg and with a body mass index between 18.5 and 24.9,
* Able and willing to participate in the research by complying with the procedures of the protocol, in particular concerning the taking of the product under study and the performance of sequential blood tests,
* Having freely signed the consent form after adequate information on the proposed study, in accordance with Good Clinical Practice and after submission of the information leaflet,
* Affiliated to a social security scheme or similar.

Exclusion Criteria:

* Smoker,
* Drug addict,
* Subject with an alcohol consumption of more than 2 glasses per day,
* Taking a drug treatment or melatonin or a product containing melatonin within 48 hours prior to a kinetics visit,
* Known organic or functional abnormality of the urinary tree,
* Any medical condition that would involve a change in melatonin metabolism:

Drug intake: Fluvoxamine, 5- or 8-methoxypsoralen, cimetidine, carbamazepine and rifampicin, analgesics, Liver abnormality known or detected at the screening visit and judged to be clinically significant by the investigator, Known autoimmune disease,

* Subject assessed as "moderately" or "definitely" evening type,
* Known hypertension (>140/90),
* Diagnosis of migraine by a health professional according to the International Headache Society (IHS) criteria revised in 2004,
* Wuth a sleep disorder,
* Thyroid dysfunction, hyperglycemia or anemia judged to be clinically significant by the investigator,
* Blood donation within one month prior to inclusion,
* A known organic or psychological abnormality (including a history of severe depression) that may bias the results of the study as judged by the investigator,
* Workers with atypical working hours (night work, staggered working hours),
* Known allergy or intolerance to any of the components of the product,
* Psychological or linguistic inability to understand and sign informed consent,
* Participant in another interventional clinical trial or during a period of exclusion from a previous clinical trial,
* Under legal protection (guardianship, curatorship) or deprived of his rights as a result of the administrative or judicial decision,
* Subject who has reached the maximum threshold for compensation for research provided for in the regulations.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
evolution of the plasma melatonin concentration | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  the change in plasma melatonin concentration

SECONDARY OUTCOMES:
evolution of the plasma concentration of 6-sulfatoxymelatonin | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  the change in plasma 6-sulfatoxymelatonin concentration
evolution of the urinary concentration of 6-sulfatoxymelatonin | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  the change in urinary 6-sulfatoxymelatonin concentration
evolution of the salivary concentration of melatonin | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  the change in salivary melatonin concentration
adverse events | during study participation, maximum 45 days
  adverse events
plasma melatonin AUC | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  Area Under the Curve of plasma melatonin
plasma 6-sulfatoxymelatonin AUC | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  Area Under the Curve of plasma 6-sulfatoxymelatonin
urinary 6-sulfatoxymelatonin AUC | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  Area Under the Curve of urinary 6-sulfatoxymelatonin
salivary melatonin AUC | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  Area Under the Curve of salivary melatonin
plasma melatonin Cmax | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  Peak concentration of plasma melatonin
plasma 6-sulfatoxymelatonin Cmax | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  Peak concentration of plasma 6-sulfatoxymelatonin
urinary 6-sulfatoxymelatonin Cmax | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  Peak concentration of urinary 6-sulfatoxymelatonin
salivary melatonin Cmax | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  Peak concentration of salivary melatonin
plasma melatonin Tmax | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  Time take to reach Cmax of plasma melatonin
plasma 6-sulfatoxymelatonin Tmax | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  Time take to reach Cmax of plasma 6-sulfatoxymelatonin
urinary 6-sulfatoxymelatonin Tmax | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  Time take to reach Cmax of urinary 6-sulfatoxymelatonin
salivary melatonin Tmax | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  Time take to reach Cmax of salivary melatonin
plasma melatonin half life | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  time required for the concentration of plasma melatonin to decrease to half of its starting dose
plasma 6-sulfatoxymelatonin half life | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  time required for the concentration of plasma 6-sulfatoxymelatonin to decrease to half of its starting dose
urinary 6-sulfatoxymelatonin half life | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  time required for the concentration of urinary 6-sulfatoxymelatonin to decrease to half of its starting dose
salivary melatonin half life | over 540 minutes after taking the sustained-release tablet and 420 minutes after taking the spray.
  time required for the concentration of salivary melatonin to decrease to half of its starting dose

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Claustrat, Study Director — PiLeJe
Locations (1):
- CIC CEN EXPERIMENTAL / CEN Nutriment, Dijon, France

IPD SHARING:
Plan to Share IPD: No
no sharing

REFERENCES:
- [Derived] Ait Abdellah S, Raverot V, Gal C, Guinobert I, Bardot V, Blondeau C, Claustrat B. Bioavailability of Melatonin after Administration of an Oral Prolonged-Release Tablet and an Immediate-Release Sublingual Spray in Healthy Male Volunteers. Drugs R D. 2023 Sep;23(3):257-265. doi: 10.1007/s40268-023-00431-9. Epub 2023 Jul 12. PMID 37438493